CLINICAL TRIAL: NCT04654364
Title: Lung Cancer Registry
Status: Recruiting | Type: Observational
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Other Study IDs: AGMT_LungCA-Reg
Record Dates: First submitted 2020-11-26; First posted 2020-12-04 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; NSCLC Stage IV; NSCLC, Stage III; SCLC, Extensive Stage; SCLC, Limited Stage
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Lung cancer is the second most common cancer in Austria with 2.868 men and 2.009 women diagnosed in 2016. Reflecting the high mortality of this disease, 2.415 men and 1.534 women died from lung cancer. Therefore, lung cancer is the most common reason for cancer associated death in men and second most common reason in women.

This malignant disease can be divided into two main groups: small cell lung cancer (SCLC) and non-small cell lung cancer (NSCLC). NSCLC is a paradigm for personalized medicine, with an increasing number of targetable gene alterations. Despite this growing diversity of molecular subtypes, in most patients no targetable mutation can be detected. For these patients check-point inhibitors with or without chemotherapy is the mainstay of the initial tumor therapy. Until recently, little progress has been made in the treatment of SCLC in last decades. Recently, an overall survival benefit by the addition of an immune-checkpoint inhibitor to first-line chemotherapy for advanced SCLC has been reported.

Despite the progress in the treatment of NSCLC, the performance of predictive biomarkers is weak. Therefore, the development of more precise prediction models is of great importance for the progress of personalized treatment strategies.

DETAILED DESCRIPTION:
This registry is designed as multicenter observational cohort of patients with lung cancer. Patient medical, testing and treatment information will be obtained through extraction of data from existing patient medical charts. Longitudinal follow-up data, including survival and tumor progression, will also be extracted from patient medical charts. This patient follow-up data will be obtained until patient death or loss to follow-up.

For documentation in the registry, no further diagnostic or therapeutic measures are required than those already necessary in general. Participation in the registry must not interfere with treatment routines. Only routine data, which has already been recorded in the patient's medical chart, is transferred to the electronic Case Report Forms. To maintain patient confidentiality, each patient will be assigned a unique patient identifying number upon enrollment; this number will accompany the patient's medical and other registry information throughout the lifetime of the registry.

A written consent must be obtained prior to the input of data. No informed consent is required from deceased patients.

Data will be collected from all sites willing to participate.

ELIGIBILITY:
Inclusion Criteria:

* stage III A-C and IV A-B NSCLC
* limited disease (LD) and extensive disease (ED) SCLC)
* patients ≥ 18 years

Exclusion Criteria:

- Due to the non-interventional design of the registry there are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry will be made available for all disciplines and physicians caring for cancer patients with locally advanced or metastatic lung cancer in Austria. In a first step patients with diagnosis after 01.01.2019 will be included. In a second step the registry will be expanded to include patients with diagnosis before 01.01.2019.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
General characteristics | 10 years
  To describe the general characteristics of advanced or metastatic stage patients in Austria (Stage III A-C and IV A-B NSCLC, limited disease (LD) and extensive disease (ED) SCLC)
Molecular testing | 10 years
  To describe molecular testing in patients with advanced or metastatic lung cancer
  * number of patients with molecular testing
  * methods for molecular testing
  * number of patients with PD-L1 testing
    * PD-L1 % range per disease stage
    * PD-L1 test antibody used
  * number of genes tested
  * number of patients with at least one mutation identified
  * number of patients with at least one druggable target identified
Characterize subgroups | 10 years
  To describe and characterize subgroups
  * Number of patients with NSCLC
  * Number of patients that receive immune-checkpoint inhibitors
  * Number of patients with targetable/druggable mutations
Treatment duration | 10 years
  To describe duration of treatment
Treatment frequency | 10 years
  To describe frequency of treatment
Degree of treatment response | 10 years
  To describe degree of treatment response in %
Treatment sequence | 10 years
  To describe sequence of use of various treatments
Outcome OS | 10 years
  To describe patient outcome by means of overall survival (OS) in %
Outcome PFS | 10 years
  To describe patient outcome by means of progression free survival (PFS) in %
Toxicity of treatment | 10 years
  To describe number of patients with toxicity of treatment with a focus on immune related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Study Chair — AGMT gemeinnützige GmbH
Locations (3):
- Austria (3):
  - Universitätsklinik für Innere Medizin III, PMU Salzburg, Salzburg, Salzburg
  - Univ.-Klinik für Innere Medizin V, Hämatologie/Onkologie LKH-Innsbruck / Universitätskliniken, Innsbruck, Tyrol
  - Kepler Universitätsklinikum GmbH, Med. Campus III, Klinik für Lungenheilkunde / Pneumologie, Linz, Upper Austria

IPD SHARING:
Plan to Share IPD: No